CLINICAL TRIAL: NCT05309993
Title: INvestigation of TENS Efficacy Versus Posterior Tibial Nerve Stimulation for Overactive Bladder
Acronym: INTENSE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate recruitment with expiration of funding and futility of enrollment
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Kate V Meriwether, MD, Assistant Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-003
Record Dates: First submitted 2022-02-25; First posted 2022-04-04 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Overactive Bladder; Overactive Bladder Syndrome; Urinary Urge Incontinence; Urinary Bladder, Overactive; Urinary Incontinence, Urge
Keywords: overactive bladder; urinary frequency; urinary urgency; urge incontinence; electrical stimulation; TENS; PTNS; nerve stimulation; bladder treatment
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Posterior Tibial Nerve Stimulation (PTNS) (Active Comparator): Women randomized to the PTNS will be scheduled for sessions once weekly for 30 minutes, for 12 weeks total. The patient sits reclined with their legs elevated on a foot rest. After alcohol swab, a 34 gauge needle is inserted percutaneously 5 cm cephalad to the medial malleolus of the right or left ankle (patient's choice) at a 60 degree angle. A surface electrode is placed on the medial ipsilateral heel. The needle and electrode are connected to a low voltage (9V) electrical stimulator. Stimulation current with a fixed frequency of 20 Hz and a pulse width of 200 μsec is increased until flexion of the big toe or fanning of all toes visualized, or until the woman reports a tingling sensation across the heel or sole of the foot. The current is then set to the highest level of tolerable to the patient (0-10 mA) and then she undergoes therapy for 30 minutes.
  Interventions: Device: PTNS
- Home transcutaneous electrical nerve stimulation (TENS) (Experimental): Women randomized to the TENS group will be asked to purchase a TENS 7000 device (estimated cost $30) and will administer self-treatment at home, daily for 20 minutes, for 12 weeks total.
  TENS treatment will be performed as follows (adapted from the most common setting from a s systematic review of TENS for OAB):
  - Surface electrodes, 2 x 2 in diameter, will be placed 5 cm cephalad to the medial malleolus of the right or left ankle (patient's choice). The second surface electrode is placed on the medial aspect of the ipsilateral calcaneus. The electrodes are connected to the TENS device with pre-set settings.
  Women will complete 20-minute daily TENS treatment for 12 weeks total.
  Interventions: Device: TENS

INTERVENTIONS:
Device: PTNS — See arm description
  Other Names: Posterior Tibial Nerve Stimulation
  Arms: Posterior Tibial Nerve Stimulation (PTNS)
Device: TENS — See arm description
  Other Names: transcutaneous electrical nerve stimulation
  Arms: Home transcutaneous electrical nerve stimulation (TENS)

SUMMARY:
The objective of this research is to perform a non-masked, non-inferiority randomized controlled trial to assess the quality of life (QOL) of women with idiopathic overactive bladder (OAB) before and after treatment with percutaneous tibial nerve stimulation (PTNS) or transcutaneous electrical nerve stimulation (TENS) of tibial nerve. The target population is patients with OAB who previously failed first- and second-line treatments and desire non-surgical management.

DETAILED DESCRIPTION:
The investigators plan to perform an unmasked, non-inferiority randomized controlled trial to determine if the quality of life is improved with the use of TENS compared to PTNS for urgency urinary incontinence and overactive bladder. Women will be informed of the arm of the study to which they are randomized, as the intervention is unable to be masked. All women will give written consent prior to enrollment.

The investigators will recruit women with OAB and/or UUI who present to the University of New Mexico Urogynecology practice at UNM Eubank Clinic (UNM) or Sandoval Regional Medical Center (SRMC) with OAB, urgency urinary incontinence (UUI) without other types of incontinence, or mixed urinary incontinence with urge predominant-symptoms who have failed a trial of at least one medication. To confirm diagnosis and eligibility, the investigators will conduct a standard intake history and physical, complete with cough stress test, POP-Q pelvic examination, urinalysis and urine culture. If the potential participant predominantly complains of OAB or UUI, she will be introduced to the study and provided with written information that may help her decide if participation in the study is right for her. All potential participants will be counseled about possible treatment options for OAB and UUI including non-surgical and surgical techniques. If a woman is withdrawn from the study either by her desire or that of the research staff, or does not desire to participate, she will be offered the same treatment options.

Recruitment will take place either in private exam rooms at these clinics or over HIPAA compliant telephone or Zoom conversation. After recruitment, they will undergo the informed consent via the same means as recruitment and complete initial questionnaires in clinic or will be sent a copy (digital or mail) to complete if enrolled virtually. Patients in the TENS group will be given their TENS device in clinic and research staff will assist in educating participants on proper placement and use of the device, as well as provide a standardized treatment protocol they will complete at home. The patients randomized to PTNS will have their sessions at the UNM Eubank Women's Primary Care Clinic.

The primary aim of the study is to determine if symptoms and quality of life related to overactive bladder are improved similarly with TENS use versus PTNS in women with OAB/UUI. If the patient is interested in non-surgical management with PTNS and fulfills study inclusion criteria, the investigators will then offer her the choice of volunteering for the study. All women will give written and/or electronic consent prior to their enrollment at this time and fill out baseline questionnaires in the clinic. Research staff and clinicians will obtain consent and administer study. After enrollment, participants will fill out a baseline OAB-q and will be given a 3-day voiding diary to complete prior to starting their intervention. Urinalysis and urine culture will be obtained to rule out urinary tract infection. This is routinely done on all new patients in the clinic and would be performed on patients not participating in the study as well. Data collected in addition to the above outcome measures includes patient demographics, medical/surgical history, and contact information, which are attached as supporting documents. This information will be collected from the patient on the day of enrollment and the investigators will review the patient's medical record if information is missing or unclear.

The randomization sequence will be generated by computer-based randomization in a sequence that preserves 1:1 randomization and also preserves allocation concealment (likely with randomly alternating block sizes of 6-10 in blocked randomization). Randomization assignments will be completed via REDCAP by a research coordinator. Randomization will only occur after consent has been signed and all baseline data has been obtained.

This is a single-center study at the University of New Mexico, and this site will recruit up to 130 patients.

Outcomes collected: Outcomes will be collected at baseline, 6 weeks, and 12 weeks, and will involve patient questionnaires such a the OAB-q (overactive bladder questionnaire), a validated tool to assess the patient's perceptions of symptom bother and impart on HRQL among patients with both continent and incontinent OAB. It is comprised of 8 symptom bother questions and 25 HRQL questions that form 4 subscales (coping, concern, sleep, and social interaction) and a total HRQL score. OAB-q is widely utilized in OAB/UUI. It will also include a voiding trial, which is a patient completed record of micturition behavior to obtain objective data on subjective symptoms. The International Continence Society (ICS) recommends use of voiding diaries in the clinical assessment of patients with lower urinary tract symptoms2. It is a chart where patients record their urinary habits for at least 24 hours and is widely used in OAB/UUI. Lastly, the study will measure the Patient Satisfaction Question (PSQ), which is a validated tool to assess patient satisfaction of treatment. It is comprised of a single question and is widely used in OAB/UUI.

Data Analysis:

Between and within group differences will be evaluated using Fisher's exact test for categorical variables and t-tests for continuous variables, as the investigators expect the data will be normally distributed. Wilcoxon rank-sum test will be used for continuous variables that are not normally distributed. If there are any baseline differences between groups, a multivariate analysis will determine the contribution of these differences to observed differences (if any) between groups.

Intention-to-treat analysis: The investigators plan to perform the primary analysis as "intention-to-treat" indicating that patients will be analyzed in the group to which they were randomized, regardless of compliance with study procedures, unless they asked to be withdrawn or were withdrawn by investigators due to safety or validity concerns. For example, PTNS patients that miss more than one session or do not make up a missed session of their office PTNS would still be analyzed in the "intention-to-treat" analysis as being in the PTNS group.

Per protocol analysis: The investigators plan to perform a secondary analysis as "per protocol" indicating that patients will be analyzed in the group to which they were randomized only if they complete a full 12 weeks of treatment in compliance with study procedures, meaning that women assigned to the PTNS arm completed 12 weekly PTNS session in the office in 13 weeks or less, and women in the at-home TENS arm performed TENS stimulation at least 5 days per week for 12 weeks, as averaged over 12 weeks. For example, PTNS patients that miss more than one session or do not make up a missed session of their office PTNS will not be analyzed in the "per protocol" analysis as being in the PTNS group.

Sample size calculation: The primary outcome for this study is the change in the OAB-q HRQOL score from baseline to 3 months. The study team used the means and standard deviation for this questionnaire from an unpublished pilot RCT study from Walter Reed that compares PTNS and TENS for the treatment of OAB (unpublished work). The investigators have powered the study based on a 10-point difference as significant between groups. This 10-point difference used for the power calculation is based on the previously established minimum important difference. To achieve power for this non-inferiority RCT study showing that the difference between groups is less than 10 points, the study will require 40 patients per group (80 total) to detect no difference with alpha = 0.05 and 80% power. Allowing for dropout of up to 30%, the investigators aim to randomize 114 patients, and will plan to recruit up to 130 to allow for potentially higher drop-out, as the study primary outcome is at the 12 weeks' time point. As the investigators plan to perform both per-protocol and intention-to-treat analysis, the sample size must be met for both per-protocol and intention-to-treat analysis, with the per-protocol patients (those in the PTNS group completing at 12 treatments in a total of 13 weeks) being expected to be a lower sample size.

Data Management/Confidentiality:

Participants will be given a de-identified study subject number. Data collection sheets and questionnaires will contain the subject number. No other patient identifiers will be collected on study forms. PHI including patient name, date of birth, phone number, email address and medical record number will be collected to track appointments and ensure patient follow-up. The data collection, HIPAA and consent forms will be maintained in a locked file cabinet in the locked Eubank research office or via REDCap. A separate folder will be designated for each participant. PHI will not be entered into the study database. The link between PHI and study IDs will be kept on a password protected computer on a secure UNM OBGYN department server.

The study database does not include sensitive information or information requiring additional protection.

Study binders will be kept in a locked cabinet in the research administrative area. In order to further ensure patient confidentiality, the identifying information will be kept separately from the numbered study files in a locked cabinet. Electronic data entry will be performed on REDCAP, using the de-identified subject study number. The electronic data and subject link will be encrypted, password protected, and stored on the secure UNM OBGYN department server. This server's electronic security is monitored / maintained by the Health Sciences Library and Informatics Center (HSLIC). A REDCAP database will be created to collect, store and manage the data. REDCAP databases are reposed securely and all data entered is de-identified. The REDCAP database is only accessible using an individual unique login and password and access is only provided to co-investigators. Access is restricted to co-investigators and research staff and will be protected using the unique REDCAP login and password provided to each co-investigator. Access to the files and REDCAP will be restricted to research personnel and Investigators and will be locked or password-protected using the unique REDCAP login and password provided to each co-investigator. The data will be stored for 6 years after completion of analysis and study closure and then will be destroyed.

A Certificate of Confidentiality will not be used to protect data from forced release. No identifying or study related data will be transported to outside locations. There will be no audio or video recordings or photographs taken.

ELIGIBILITY:
Inclusion Criteria:

* Female Subjects ≥18 years of age
* OAB, UUI or Mixed Urinary Incontinence with urgency predominant symptoms and more bother from UUI than stress urinary incontinence
* Failed trial of conservative therapy (including bladder training, fluid modification, diet modification, caffeine restriction, or pelvic floor training) -Failed trial of at least one pharmacologic treatment (anticholinergics, β3- adrenoceptor agonist) either due to inability to take the medication, adverse reaction to medication, or no improvement on medication
* Willing to complete study questionnaires
* Willing to adhere to 12 office visits for PTNS over 3 months if randomized to that arm
* No contraindication to undergoing PTNS or TENS therapy

Exclusion Criteria:

* Age < 18 years
* Presence of urinary fistula
* Male genital anatomy
* Undergoing evaluation or treatment of recurrent (2 or more infections in the last 6 months or 3 or more infections in the last 12 months) or current urinary tract infection
* Current Bladder stones
* Bladder cancer or suspected bladder cancer
* Gross Hematuria
* Pregnancy or planning to become pregnant during the study
* Cognitive impairment
* Central or peripheral neurologic disorders such as multiple sclerosis, Parkinson's disease, spina bifida, spinal cord lesions, etc.
* Metal implants such as pacemaker, implantable defibrillator, or metal implants where PTNS or TENS device needs to be placed (ankle/leg)
* Uncontrolled diabetes
* Diabetes with peripheral nerve involvement
* Current use of anticoagulants (excluding aspirin)
* Current use of anticholinergics or use within the last 4 weeks
* Current use of botox bladder injections or bladder botox injection within the last year (12 months)
* Current use of sacral neuromodulation therapy or currently implanted sacral neuromodulation device or leads
* Bladder outlet obstruction
* Urinary retention or gastric retention
* Painful Bladder Syndrome/Interstitial Cystitis
* Unable to be contacted for follow up by telephone
* Inability to speak/read/understand English or Spanish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females are entered in this trial as they are population most affected by overactive bladder (OAB) and served by the investigators
Enrollment: 27 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Overactive bladder Questionnaire (OAB-q) Health-Related Quality of Life (HRQOL) score | 12 weeks
  Change in OAB-q HRQOL score from baseline to 12 weeks, score range 0 to 100, higher scores indicating higher quality of life (higher scores good)

SECONDARY OUTCOMES:
Overactive bladder questionnaire (OAB-q) Symptom Bother subscale score | 6 weeks, 12 weeks
  OAB-q Symptom Bother subscale score change from baseline to time point, scores ranging from 0 to 100, higher scores indicating higher bother/worse symptoms (higher scores bad)
Overactive bladder Questionnaire (OAB-q) Health-Related Quality of Life | 6 weeks
  Change in OAB-q HRQOL score from baseline to 12 weeks, score range 0 to 100, higher scores indicating higher quality of life (higher scores good)
Number of urinary incontinence episodes | 6 weeks, 12 weeks
  Number of urinary incontinence episodes on 3-day voiding diary
Number of voids per day | 6 weeks, 12 weeks
  Number of voids per day on 3-day voiding diary
Number of voids per night | 6 weeks, 12 weeks
  Number of voids per night on 3-day voiding diary
Patient satisfaction question (PSQ) | 6 weeks, 12 weeks
  Patient satisfaction question is a single question asking: "How satisfied are you with your progress in this program?", where patients answer on a Likert scale the possible responses of "completely", "somewhat", and "not at all".
Patient compliance | 6 weeks, 12 weeks
  Number of treatment sessions completed
Adverse events | Weekly for 12 weeks
  Adverse events reported during research

CONTACTS AND LOCATIONS:
Overall Officials: Kate V Meriwether, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gopal M, Haynes K, Bellamy SL, Arya LA. Discontinuation rates of anticholinergic medications used for the treatment of lower urinary tract symptoms. Obstet Gynecol. 2008 Dec;112(6):1311-1318. doi: 10.1097/AOG.0b013e31818e8aa4. PMID 19037041
- [Background] Monga AK, Tracey MR, Subbaroyan J. A systematic review of clinical studies of electrical stimulation for treatment of lower urinary tract dysfunction. Int Urogynecol J. 2012 Aug;23(8):993-1005. doi: 10.1007/s00192-012-1691-5. Epub 2012 Mar 17. PMID 22426872
- [Background] Lightner DJ, Gomelsky A, Souter L, Vasavada SP. Diagnosis and Treatment of Overactive Bladder (Non-Neurogenic) in Adults: AUA/SUFU Guideline Amendment 2019. J Urol. 2019 Sep;202(3):558-563. doi: 10.1097/JU.0000000000000309. Epub 2019 Aug 8. PMID 31039103
- [Background] Sutherland SE, Lavers A, Carlson A, Holtz C, Kesha J, Siegel SW. Sacral nerve stimulation for voiding dysfunction: One institution's 11-year experience. Neurourol Urodyn. 2007;26(1):19-28; discussion 36. doi: 10.1002/nau.20345. PMID 17078071
- [Background] Kraus SR, Shiozawa A, Szabo SM, Qian C, Rogula B, Hairston J. Treatment patterns and costs among patients with OAB treated with combination oral therapy, sacral nerve stimulation, percutaneous tibial nerve stimulation, or onabotulinumtoxinA in the United States. Neurourol Urodyn. 2020 Nov;39(8):2206-2222. doi: 10.1002/nau.24474. Epub 2020 Aug 22. PMID 32827230
- [Background] Peters KM, Carrico DJ, Perez-Marrero RA, Khan AU, Wooldridge LS, Davis GL, Macdiarmid SA. Randomized trial of percutaneous tibial nerve stimulation versus Sham efficacy in the treatment of overactive bladder syndrome: results from the SUmiT trial. J Urol. 2010 Apr;183(4):1438-43. doi: 10.1016/j.juro.2009.12.036. Epub 2010 Feb 20. PMID 20171677
- [Background] Peters KM, Carrico DJ, MacDiarmid SA, Wooldridge LS, Khan AU, McCoy CE, Franco N, Bennett JB. Sustained therapeutic effects of percutaneous tibial nerve stimulation: 24-month results of the STEP study. Neurourol Urodyn. 2013 Jan;32(1):24-9. doi: 10.1002/nau.22266. Epub 2012 Jun 5. PMID 22674493
- [Background] Staskin DR, Peters KM, MacDiarmid S, Shore N, de Groat WC. Percutaneous tibial nerve stimulation: a clinically and cost effective addition to the overactive bladder algorithm of care. Curr Urol Rep. 2012 Oct;13(5):327-34. doi: 10.1007/s11934-012-0274-9. PMID 22893501
- [Background] Peters KM, Macdiarmid SA, Wooldridge LS, Leong FC, Shobeiri SA, Rovner ES, Siegel SW, Tate SB, Jarnagin BK, Rosenblatt PL, Feagins BA. Randomized trial of percutaneous tibial nerve stimulation versus extended-release tolterodine: results from the overactive bladder innovative therapy trial. J Urol. 2009 Sep;182(3):1055-61. doi: 10.1016/j.juro.2009.05.045. Epub 2009 Jul 18. PMID 19616802
- [Background] MacDiarmid SA, Peters KM, Shobeiri SA, Wooldridge LS, Rovner ES, Leong FC, Siegel SW, Tate SB, Feagins BA. Long-term durability of percutaneous tibial nerve stimulation for the treatment of overactive bladder. J Urol. 2010 Jan;183(1):234-40. doi: 10.1016/j.juro.2009.08.160. PMID 19913821
- [Background] Burton C, Sajja A, Latthe PM. Effectiveness of percutaneous posterior tibial nerve stimulation for overactive bladder: a systematic review and meta-analysis. Neurourol Urodyn. 2012 Nov;31(8):1206-16. doi: 10.1002/nau.22251. Epub 2012 May 11. PMID 22581511
- [Background] Schreiner L, dos Santos TG, Knorst MR, da Silva Filho IG. Randomized trial of transcutaneous tibial nerve stimulation to treat urge urinary incontinence in older women. Int Urogynecol J. 2010 Sep;21(9):1065-70. doi: 10.1007/s00192-010-1165-6. Epub 2010 May 11. PMID 20458465
- [Background] Schreiner L, Nygaard CC, Dos Santos TG, Knorst MR, da Silva Filho IG. Transcutaneous tibial nerve stimulation to treat urgency urinary incontinence in older women: 12-month follow-up of a randomized controlled trial. Int Urogynecol J. 2021 Mar;32(3):687-693. doi: 10.1007/s00192-020-04560-6. Epub 2020 Oct 15. PMID 33057739
- [Background] Booth J, Connelly L, Dickson S, Duncan F, Lawrence M. The effectiveness of transcutaneous tibial nerve stimulation (TTNS) for adults with overactive bladder syndrome: A systematic review. Neurourol Urodyn. 2018 Feb;37(2):528-541. doi: 10.1002/nau.23351. Epub 2017 Jul 21. PMID 28731583
- [Background] Daly CME, Loi L, Booth J, Saidan D, Guerrero K, Tyagi V. Self-management of overactive bladder at home using transcutaneous tibial nerve stimulation: a qualitative study of women's experiences. BMC Womens Health. 2021 Oct 27;21(1):374. doi: 10.1186/s12905-021-01522-y. PMID 34706709
- [Background] Ramirez-Garcia I, Blanco-Ratto L, Kauffmann S, Carralero-Martinez A, Sanchez E. Efficacy of transcutaneous stimulation of the posterior tibial nerve compared to percutaneous stimulation in idiopathic overactive bladder syndrome: Randomized control trial. Neurourol Urodyn. 2019 Jan;38(1):261-268. doi: 10.1002/nau.23843. Epub 2018 Oct 12. PMID 30311692
- [Background] Coyne KS, Matza LS, Thompson CL, Kopp ZS, Khullar V. Determining the importance of change in the overactive bladder questionnaire. J Urol. 2006 Aug;176(2):627-32; discussion 632. doi: 10.1016/j.juro.2006.03.088. PMID 16813906
- [Background] Dyer KY, Xu Y, Brubaker L, Nygaard I, Markland A, Rahn D, Chai TC, Stoddard A, Lukacz E; Urinary Incontinence Treatment Network (UITN). Minimum important difference for validated instruments in women with urge incontinence. Neurourol Urodyn. 2011 Sep;30(7):1319-24. doi: 10.1002/nau.21028. Epub 2011 May 11. PMID 21563210
- [Background] Coyne KS, Matza LS, Thompson CL. The responsiveness of the Overactive Bladder Questionnaire (OAB-q). Qual Life Res. 2005 Apr;14(3):849-55. doi: 10.1007/s11136-004-0706-1. PMID 16022077
- [Background] Coyne K, Revicki D, Hunt T, Corey R, Stewart W, Bentkover J, Kurth H, Abrams P. Psychometric validation of an overactive bladder symptom and health-related quality of life questionnaire: the OAB-q. Qual Life Res. 2002 Sep;11(6):563-74. doi: 10.1023/a:1016370925601. PMID 12206577
- [Background] Matza LS, Thompson CL, Krasnow J, Brewster-Jordan J, Zyczynski T, Coyne KS. Test-retest reliability of four questionnaires for patients with overactive bladder: the overactive bladder questionnaire (OAB-q), patient perception of bladder condition (PPBC), urgency questionnaire (UQ), and the primary OAB symptom questionnaire (POSQ). Neurourol Urodyn. 2005;24(3):215-25. doi: 10.1002/nau.20110. PMID 15747340
- [Background] Salatzki J, Liechti MD, Spanudakis E, Gonzales G, Baldwin J, Haslam C, Pakzad M, Panicker JN. Factors influencing return for maintenance treatment with percutaneous tibial nerve stimulation for the management of the overactive bladder. BJU Int. 2019 May;123(5A):E20-E28. doi: 10.1111/bju.14651. Epub 2019 Feb 3. PMID 30552801
- [Background] van der Pal F, van Balken MR, Heesakkers JP, Debruyne FM, Bemelmans BL. Percutaneous tibial nerve stimulation in the treatment of refractory overactive bladder syndrome: is maintenance treatment necessary? BJU Int. 2006 Mar;97(3):547-50. doi: 10.1111/j.1464-410X.2006.06055.x. PMID 16469023
- [Background] Locher JL, Goode PS, Roth DL, Worrell RL, Burgio KL. Reliability assessment of the bladder diary for urinary incontinence in older women. J Gerontol A Biol Sci Med Sci. 2001 Jan;56(1):M32-5. doi: 10.1093/gerona/56.1.m32. PMID 11193230
- [Background] de Seze M, Raibaut P, Gallien P, Even-Schneider A, Denys P, Bonniaud V, Game X, Amarenco G. Transcutaneous posterior tibial nerve stimulation for treatment of the overactive bladder syndrome in multiple sclerosis: results of a multicenter prospective study. Neurourol Urodyn. 2011 Mar;30(3):306-11. doi: 10.1002/nau.20958. Epub 2011 Feb 8. PMID 21305588
- [Background] Bright E, Drake MJ, Abrams P. Urinary diaries: evidence for the development and validation of diary content, format, and duration. Neurourol Urodyn. 2011 Mar;30(3):348-52. doi: 10.1002/nau.20994. Epub 2011 Jan 31. PMID 21284023
- [Background] Burgio KL, Goode PS, Richter HE, Locher JL, Roth DL. Global ratings of patient satisfaction and perceptions of improvement with treatment for urinary incontinence: validation of three global patient ratings. Neurourol Urodyn. 2006;25(5):411-7. doi: 10.1002/nau.20243. PMID 16652380
- [Background] Goode PS, Burgio KL, Kraus SR, Kenton K, Litman HJ, Richter HE; Urinary Incontinence Treatment Network. Correlates and predictors of patient satisfaction with drug therapy and combined drug therapy and behavioral training for urgency urinary incontinence in women. Int Urogynecol J. 2011 Mar;22(3):327-34. doi: 10.1007/s00192-010-1287-x. Epub 2010 Oct 13. PMID 20945064
- [Background] Ammi M, Chautard D, Brassart E, Culty T, Azzouzi AR, Bigot P. Transcutaneous posterior tibial nerve stimulation: evaluation of a therapeutic option in the management of anticholinergic refractory overactive bladder. Int Urogynecol J. 2014 Aug;25(8):1065-9. doi: 10.1007/s00192-014-2359-0. Epub 2014 Mar 6. PMID 24599180

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT05309993/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT05309993/ICF_001.pdf